CLINICAL TRIAL: NCT00459966
Title: Preoperative Prevention and Early Rehabilitation for Patients Undergoing Elective Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01-041/03
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2007-04

CONDITIONS: Spine Surgery
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Preoperative rehabilitation

SUMMARY:
Aim: The aim is to evaluate the outcome after spine surgery when using an integrated program that combined preoperative prevention and early postoperative rehabilitation compared to the routine procedures.

Outcome measurements: Postoperative hospital stay, complications, function, pain, and patient satisfaction.

Method: 60 patients scheduled for surgery for degenerative lumbar disease. The control group followed the routines in the department. The intervention group followed the integrated program consisting of preoperative prevention.

DETAILED DESCRIPTION:
Introduction: An increasing number of patients undergo surgery for degenerative spine disease, which is, however, related to a significant development of postoperative complications. Evidence has been gathered for other surgical procedures about improved outcome after early rehabilitation programs (fast track surgery), preoperative smoking and alcohol cessation programs, respectively. Hitherto, no studies have been published concerning a combined program of the preoperative prevention programs and fast track surgery.

Aim: The aim is to evaluate the outcome after spine surgery when using an integrated program that combined preoperative prevention and early postoperative rehabilitation compared to the routine procedures.

Outcome measurements: Postoperative hospital stay, complications, function, pain, and patient satisfaction.

Method: 60 patients scheduled for surgery for degenerative lumbar disease were computer-randomized to intervention. The control group followed the routines in the department. The intervention group followed the integrated program consisting of preoperative prevention, which began 2 months prior to the operation: an exercise program designed to strengthen the muscles of the spine, and optimization of the analgetic treatment. Smokers and harmful drinkers were offered cessation intervention. The day before surgery all had enteral protein supplement.

Early postoperative rehabilitation included balanced pain therapy, including self-administered epidural analgesia, intensified mobilization immediately after surgery and enteral protein supplement.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative lumbar disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-02; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Per Rotboell Nielsen, MD, Principal Investigator — uaffiliatation
Locations (1):
- Head-Ortho-Centre, Anesthesiology Department, Rigshospitalet,, Copenhagen, Denmark